CLINICAL TRIAL: NCT03139851
Title: CHEMOIMMUNE - A Phase II Study Evaluating an Anti-PD1 Monoclonal Antibody (Pembrolizumab) in Lymphopenic Metastatic Breast Cancer Patients Treated With Metronomic Cyclophosphamide
Brief Title: Evaluation of Pembrolizumab in Lymphopenic Metastatic Breast Cancer Patients Treated With Metronomic Cyclophosphamide
Acronym: CHEMOIMMUNE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET16-073; 2016-002736-33 (EudraCT Number)
Record Dates: First submitted 2017-04-10; First posted 2017-05-04 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2020-08

CONDITIONS: Metastatic Breast Cancer
Keywords: Solid tumor; Breast cancer; Metastatic cancer; Pembrolizumab; Metronomic cyclophosphamide
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Cyclophosphamide; pembrolizumab; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cyclophosphamide and Pembrolizumab (Other): The treatments received are:
  * cyclophosphamide (50 mg/day, daily, per os)
  * pembrolizumab (200 mg every 3 weeks, intravenously [IV]). On days 1, cyclophosphamide should be taken first and pembrolizumab infusion initiated within 1 hour after cyclophosphamide intake.
  Interventions: Drug: Cyclophosphamide 50mg; Drug: Pembrolizumab 100 MG in 4 ML Injection

INTERVENTIONS:
Drug: Cyclophosphamide 50mg — One tablet per day. Cyclophosphamide will continue to be administered as long as patient experiences clinical benefit in the opinion of the investigator or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.
Drug: Pembrolizumab 100 MG in 4 ML Injection — IV infusion every 3 weeks. Pembrolizumab will continue to be administered as long as patient experiences clinical benefit in the opinion of the investigator or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.
  Other Names: Keytruda

SUMMARY:
The investigators hypothesize that the administration of pembrolizumab combined to metronomic cyclophosphamide may be an interesting therapeutic option for female patients breast cancer with lymphopenia.

Include only patients with breast cancer with lymphopenia is based on the particularly poor prognosis of these patients. The approach suggested here is to deplete and active the immune response of these immunosuppressed patients. The combination of pembrolizumab and cyclophosphamide would provide a higher gain in anti-tumor response in these patients than in those without lymphopenia and in chemotherapy alone.

The investigators proposal is to conduct a multicentric, non-comparative, single arm, two-stage, Phase II trial in lymphopenic patients with metastatic breast cancer.

The study is divided in 2 parts:

* a safety run-in Phase aiming to evaluate the safety of the combination therapy pembrolizumab + metronomic cyclophosphamide based on the occurrence of severe toxicities.
* a two-stage Phase II aiming to evaluate the clinical activity of the combination therapy pembrolizumab + metronomic cyclophosphamide.

In both parts of the study, patients will receive cyclophosphamide (50 mg/day, daily, per os) and pembrolizumab (200 mg every 3 weeks, intravenously [IV]). The adverse events of the two drugs are well known.

DETAILED DESCRIPTION:
The initiation of different stage of the study depend on the occurrences of severe toxicities in safety run-in phase and Clinical Benefit rate after 24 weeks in the two-stage Phase II of the study.

Both study drugs will continue to be administered as long as patient experience clinical benefit in the opinion of the investigator or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Female patient>=18 years of age on day of signing informed consent.
* Histologically proven HER2-negative metastatic breast cancer. HER2-negativity is defined as immunohistochemistry (IHC) score 0, 1+ or 2+ and fluorescent in situ hybridization (FISH) negative or just FISH negative, whichever was performed.
* Patient previously treated with at least one prior line of standard chemotherapy either in the adjuvant setting or in the metastatic setting. Patients may be included in the first line metastatic setting if they have received anthracycline and/or taxane-based therapy in the neoadjuvant/adjuvant setting.

Note: Patients with ER-positive tumors must have received at least one prior endocrine therapy, either in the adjuvant setting or in the metastatic setting.

* Documented lymphopenia defined by at least one value of lymphocyte count < 1.5 G/L within 15 days before treatment start (C1D1) and following at least 15 days since the last administration of chemotherapy.
* Biopsiable disease i.e. at least one lesion with a diameter ≥ 10 mm, visible by medical imaging and accessible to percutaneous sampling.
* Patient willing to undergo 2 tumor biopsies (at inclusion and at C3D1).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1 or 2 and minimum life expectancy of 24 weeks.
* Documented radiological disease progression at time of study entry.
* At least one measurable lesion according to RECIST 1.1.
* Adequate end organ and marrow function as defined below: all screening labs should be performed within 3 days before treatment start (C1D1).

Hematological Laboratory Values Absolute neutrophil count (ANC) ≥ 1.5G/L Platelets ≥ 100G/L Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L (without transfusion within 7 days of assessment) Renal Laboratory Values Serum creatinine ≤ 1.5 X upper limit of normal (ULN) or Calculated creatinine clearance as per MDRD or CKD-EPI formula ≥ 60 mL/min /1.73m2 Hepatic Laboratory Values Serum total bilirubin ≤ 1.5 X ULN or Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN (up to 5 ULN may be tolerated in case of liver metastasis) Albumin ≥ 25 g/L Coagulation Laboratory Values International Normalized Ratio (INR) ≤ 1.5 ULN Ratio of activated Partial Thromboplastin Time (aPTT) ≤ 1.5 ULN

* Absence of prior significant treatment-related toxicity i.e. treatment-related toxicity > Grade 1 as per CTCAE v4.03, except grade 2 alopecia, grade 2 neuropathy and biological values as described in I10.
* Women of child-bearing potential must have a negative serum pregnancy test within 3 days before C1D1.
* Women of child-bearing potential must agree to use 2 effective forms of contraception from the time of the negative pregnancy test up to 120 days after the last dose of study drugs.
* Patient should understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be covered by a medical insurance.

Exclusion Criteria:

* Previously treated with more than 3 prior lines of chemotherapy in the metastatic setting
* Has previously received therapy with an anti-programmed cell death 1 (PD-1), anti-programmed cell death 1 ligand 1(PD-L1), anti-PD-L2, anti-CD137 antibody, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody.
* Presenting any contraindication to cyclophosphamide treatment including known hypersensitivity to cyclophosphamide, inflammation of the bladder (cystitis), urinary outflow obstruction or active infection.
* Requiring the use of concomitant medications defined as forbidden in the SPC of cyclophosphamide.
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has a known history of active Bacillus Tuberculosis.
* Prior treatment with:

  * any investigational agent within 4 weeks before C1D1 (or 5 half-lives whichever is shorter with a minimum of 2 weeks);
  * any systemic corticosteroids at doses higher than 10 mg/d of prednisolone or equivalent or immunosuppressive agent within 4 weeks before C1D1;
  * any monoclonal antibody within 4 weeks before C1D1;
  * any chemotherapy, targeted small molecule therapy, radiation therapy, or surgery within 2 weeks prior to C1D1.

Note: If a patient underwent a major surgical procedure, they must have adequately recovered from the toxicity (i.e. wound healing) and/or complications from the intervention prior to starting therapy.

* any live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to C1D1 and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 28 days prior to C1D1. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids at doses higher than 10 mg/d of methylprednisolone or equivalent or immunosuppressive agents.

Note: Patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Patients with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.

* Has an history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) or active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Severe Toxicities (ST) in Run-In Phase Part | First 6 weeks of treatment
  Number of severe toxicities occurring during the first 6 weeks of treatment and defined as following events evaluated as related to study drugs, using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) V4.03:
  * any Grade ≥ 3 non hematological toxicity including in particular events of special interest
  * any Grade ≥4 hematological and non-hematological Adverse Event (AE) including.
24-week Clinical Benefit Rate (CBR24w) in Phase II part | 24 weeks of treatment
  CBR24w, defined as the percentage of Complete Response (CR), (Partial Response) PR or prolonged Stable Disease (SD) i.e. SD lasting ≥ 24 weeks (pSD) within the evaluable population of patient. Response will be evaluated by Response Evaluation Criteria In Solid Tumors (RECIST) V1.1 and the CBR24w will be summarized by a proportion together with its 95% confidence interval.

SECONDARY OUTCOMES:
Overall response Rate (ORR) at 24 weeks | 24 weeks of treatment
  The objective response rate (ORR) will be defined as the proportion of patients (described on the efficacy-evaluable population) who achieve complete response (CR) or partial response (PR) as best overall response at 24 weeks of treatment. ORR is based on tumor assessments. Response will be evaluated by Response Evaluation Criteria In Solid Tumors (RECIST) V1.1
Duration of response (DoR) | 15 months
  Calculated from date of first documented objective response (i.e., CR or PR) until date of first documented progression disease.
Progression-Free Survival (PFS) | 15 months
  Measured from the date of study drugs start to the date of the first objective disease progression or death.
Overall Survival (OS) | 15 months
  Defined as the duration of time from start of treatment to time of death.
Adverse events reporting | 15 months
  Adverse Events (AE), vital signs, ECG, physical examination, laboratory safety assessments (hematological and biochemical parameters).

CONTACTS AND LOCATIONS:
Overall Officials: Olivier TREDAN, MD, Principal Investigator — Centre Leon Berard
Locations (5):
- France (5):
  - ICO - Paul Papin, Angers
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - ICO - René Gauducheau, Saint-Herblain
  - Institut de cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No